CLINICAL TRIAL: NCT01700179
Title: A Phase 1b, Open-label, Pilot Study to Evaluate the Safety, Tolerability, and Antiviral Activity of Oral ACH-0143102 Administered in Combination With Ribavirin for 12 Weeks in Treatment-naive Subjects With Chronic Hepatitis C Virus Infection Genotype 1b
Brief Title: Evaluation of Safety, Tolerability, and Antiviral Activity of ACH-0143102 Plus Ribavirin In Treatment-naive Hepatitis C Virus Infection Genotype 1b Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH102-005
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACH-0143102 plus ribavirin daily (Experimental): ACH-0143102 loading dose (225 milligrams [mg]) on Day 1, followed by maintenance doses (75 mg) on Days 2-84, plus weight-based ribavirin as per label on Days 1-84.
  Interventions: Drug: ACH-0143102; Drug: Ribavirin

INTERVENTIONS:
Drug: ACH-0143102
Drug: Ribavirin

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and efficacy of 12 weeks of treatment with ACH-0143102 and ribavirin in genotype 1b (GT1b), treatment-naive, hepatitis C virus (HCV) participants.

DETAILED DESCRIPTION:
A Phase 1b, pilot study that evaluated the safety, tolerability, and antiviral activity of oral ACH-0143102 administered in combination with ribavirin for 12 weeks in treatment-naive participants with chronic HCV GT1b.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years and older.
* Clinical diagnosis of hepatitis C with GT1b.
* Chronic hepatitis C treatment-naive participants.
* Interleukin 28B genotype CC.
* HCV ribonucleic acid > 10,000 international units/milliliter at screening.
* Female participants must be willing to use 2 effective methods of contraception during the dosing period and for 6 months after the last dose of ribavirin.
* Male participants must be willing to use an effective barrier method of contraception throughout the dosing period and for 6 months after the last dose of ribavirin. Male participants must agree not to donate sperm while enrolled in the study and for 6 months after the last dose of ribavirin.
* Willing to participate in all study activities and all study requirements.

Exclusion Criteria:

* Body mass index > 36 kilograms/meter squared.
* Pregnant or nursing females.
* Clinically significant laboratory abnormalities at screening.
* Previous participation in a clinical trial with protease inhibitor and/or non-structural protein 5A inhibitor.
* Human immunodeficiency virus infection or other liver diseases.
* Positive hepatitis B surface antigen.
* Liver cirrhosis.
* Uncontrolled psychiatric disease.
* Clinical evidence of chronic cardiac disease.
* History of malignancy of any organ system within 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 sites in the United States between 05 September 2012 and 11 December, 2012.
Pre-assignment Details: Participants were screened within 4 weeks (-28 to -1 days) before administration of the study drug. Participants who meet all eligibility criteria were instructed to arrive at the study center on the baseline day.
Groups:
- ACH-0143102 Plus Ribavirin: ACH-0143102 (225 milligrams [mg]) loading dose on Day 1, followed by maintenance doses (75 mg) on Days 2-84, plus weight-based ribavirin as per label on Days 1-84.
Period: Overall Study
Arm/Group | ACH-0143102 Plus Ribavirin
Started | 8
Completed | 6
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: The analysis population for baseline characteristics was all enrolled participants.
Groups:
- ACH-0143102 Plus Ribavirin: ACH-0143102 (225 mg) loading dose on Day 1, followed by maintenance doses (75 mg) on Days 2-84, plus weight-based ribavirin as per label on Days 1-84.
Arm/Group | ACH-0143102 Plus Ribavirin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.07 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meter squared] | 28.13 (4.183)

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response At 12 Weeks (SVR12)
Description: To determine the incidence of the SVR12 after the completion of dosing with ACH-0143102 plus ribavirin, reported as hepatitis C virus ribonucleic acid less than the limit of quantification at that time point.
Time Frame: 12 weeks following the last dose
Measure: Number; unit: percentage of participants
Arm/Group | ACH-0143102 Plus Ribavirin
Number analyzed (Participants) | 8
percentage of participants | 50

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment into the study through end of treatment plus 24 weeks of follow-up, for up to 36 weeks.
Description: Treatment-emergent adverse events are summarized.
Arm/Group | ACH-0143102 Plus Ribavirin
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ACH-0143102 Plus Ribavirin (N=8)
Anaemia (Blood and lymphatic system disorders) | 4
Atrioventricular block second degree (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Influenza like illness (General disorders) | 1
Irritability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Folliculitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Emotional disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Breast tenderness (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting/presenting a manuscript or materials relating to a Study to a publisher, reviewer, or outside person, the Institution shall provide to Sponsor a copy of all such manuscripts or materials, and Sponsor shall have thirty (30) days to review and comment. The Institution shall, upon Sponsor's request, further delay publication or presentation for a period of up to sixty (60) days to allow Sponsor to protect its interests in any Sponsor Inventions.